CLINICAL TRIAL: NCT02182804
Title: Diagnostic Values of Probe-based Confocal Laser Endomicroscopy (pCLE) and Magnifying Narrow Band Imaging (M-NBI) for Early Neoplasms Detection in Esophageal Lugol'S-voiding Lesions.
Brief Title: A Diagnostic Study of the Advanced Endoscopy to Detect Early Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Gastroenterologist, King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP008
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Neoplasms
Keywords: Confocal Laser Endomicroscopy; Narrow Band Imaging; Lugol Chromoendoscopy; Esophageal Neoplasm; Head and Neck Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Study (Experimental): probe-based confocal laser endomicroscopy narrow band imaging with magnification
  Interventions: Device: Olympus; Device: Cellvizio

INTERVENTIONS:
Device: Olympus — narrow band imaging with magnification
Device: Cellvizio — probe-based confocal laser endomicroscopy

SUMMARY:
This descriptive cross sectional study aims to directly compare the diagnostic capability of the probed-based confocal laser endomicroscopy (pCLE) and the magnifying narrow band imaging (M-NBI) in the Lugol's voiding lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 20 years
* Having histological-confirmed diagnosis of head and neck cancer
* Having no esophageal symptoms

Exclusion Criteria:

* Having index cancer of nasopharynx
* History of esophageal surgery
* Having esophageal stricture or obstruction
* Having esophageal varices
* Known case of esophageal cancer
* Uncorrectable coagulopathy and thrombocytopenia
* Pregnancy
* Thyrotoxicosis
* Creatinine clearance less than 30 ml/min
* Allergy to iodine or fluorescein.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, M.D., Principal Investigator — King Chulalongkorn Memorial Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 631 patients with a previous history of head and neck cancer in the 10-year record. Of the 631 patients, 587 were excluded for the following reasons: patients could not be contacted (n=458), death (n=72), esophageal obstruction or stricture, previous esophageal surgery (n=34), and patients who refused to participate (n=23).
Groups:
- Study Arm: Probe-based confocal laser endomicroscopy and narrow band imaging with magnification in esophageal Lugol's voiding lesions.
Period: Overall Study
Arm/Group | Study Arm
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 44

OUTCOME MEASURES:

1. Primary Outcome: Accuracy
Description: Diagnostic performance of the pCLE and M-NBI in Lugol's voiding lesions size larger than 5 millimeters.
Time Frame: an expected average of 2 weeks
Population: Twenty-one Lugol's voiding lesions larger than 5mm were detected in 12 patients.
Measure: Number (95% Confidence Interval); unit: Percentage of accuracy
Units Other Than Participants: Lugol's voiding lesion
Arm/Group | Study Arm
Number analyzed (Participants) | 12
Number analyzed (Lugol's voiding lesion) | 21
Percentage of accuracy
  pCLE | 89 [67 to 97]
  dNBI | 70 [48 to 85]

ADVERSE EVENTS:
Time Frame: Intraprocedural.
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 1/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=44)
Bleeding (Surgical and medical procedures) | 1 (1) — One patient developed bleeding after biopsy and was successfully treated with endoscopic clipping.

LIMITATIONS AND CAVEATS:
This was a pilot study and the sample size was small. We did not randomly assign the order of dNBI and pCLE. The unwashed Lugol's stain significantly influenced the observation of IPCL structure on dNBI study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No